CLINICAL TRIAL: NCT05517304
Title: Transcutaneous Vagal Nerve Stimulation in Veterans With Posttraumatic Stress Disorder
Acronym: VNS in PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHBP-004-21F; I01CX002331 (NIH)
Record Dates: First submitted 2022-08-15; First posted 2022-08-26 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Stress Disorders, Post-Traumatic; PTSD; Vagus Nerve
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: tcVNS versus sham stimulation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: sham stimulation comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- tcVNS (Experimental): Stimulation twice daily with transcutaneous Vagal Nerve Stimulation (tcVNS)
  Interventions: Device: tcVNS
- sham (Active Comparator): stimulation with sham
  Interventions: Device: sham

INTERVENTIONS:
Device: tcVNS — active stimulation with transcutaneous Vagal Nerve Stimulation (tcVNS)
  Arms: tcVNS
Device: sham — sham stimulation
  Arms: sham

SUMMARY:
This study effects the effects of transcutaneous cervical vagal nerve stimulation (tcVNS) or a sham control on brain, physiology, and PTSD symptoms in Veterans with posttraumatic stress disorder (PTSD). Veterans undergo brain imaging and physiological measures in conjunction with traumatic scripts before and after three months of twice daily treatment with tcVNS or sham stimulation at home.

DETAILED DESCRIPTION:
Description: This study assesses brain function measured with High Resolution Positron Emission Tomography (HR-PET) during exposure to stressful traumatic scripts paired with tcVNS or sham stimulation, with secondary measures of blood inflammatory biomarkers, and sympathetic function. Participants then undergo three months of twice daily home treatment with repeat measures.

Drug/Device Handling: [O-15] radiolabeled water has a half-life of 110 seconds and is made on site at the Emory Center for Systems Imaging (CSI). Dr. Bremner holds the Investigational New Drug (IND) approval for use of radiolabeled water at Emory University. The investigators have performed hundreds of studies in human subjects at Emory and there have been no adverse events or untoward effects to date.

tcVNS with the GammaCore device is approved by the Emory IRB for a recently completed study in PTSD and others in progress for Opioid Use Disorder and was shown to be well tolerated and there have been no adverse events or untoward effects with the device. The FDA granted Breakthrough Device Designation for PTSD for the gammaCore tcVNS device based on the investigators' studies. Devices are blinded by ElectroCore and the devices and information are kept by the Data Manager under double lock and key. Device records are kept by the Data Manager and stored on Redcap or secured research drives. Devices are given to the study team along with a device schedule under direct supervision from the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Veterans between the ages of 18 and 75 will be included with a diagnosis of PTSD based on DSM-5 criteria

Exclusion Criteria:

Subjects will be excluded with:

* a history of mild traumatic brain injury (mTBI) based on VA Criteria
* moderate or greater TBI
* positive pregnancy test
* meningitis or other neurological disorder
* alcohol or substance abuse use disorder based on DSM-5 criteria within the past 12 months
* current or lifetime history of schizophrenia, schizoaffective disorder, bipolar I disorder, anorexia nervosa or bulimia, based on DSM-5
* active suicidal ideation with a plan
* a history of serious medical or neurological illness, such as cardiovascular, gastrointestinal, hepatic, renal, neurologic or other systemic illness that would preclude participation based on clinical judgment of the PI
* active opiate or benzodiazepine treatment
* history of structural abnormality on brain MRI or CT if one has been performed in the past

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-11-17 (Estimated)

PRIMARY OUTCOMES:
Change in PTSD symptoms | Baseline to three months
  Change in PTSD symptoms measured with the Clinician Administered PTSD Scale (CAPS) and PTSD Checklist (PCL) in tcVNS versus sham conditions
brain | baseline
  change in brain activation in insula measured with PET in response to trauma scripts with VNS compared to sham

SECONDARY OUTCOMES:
sympathetic function | baseline
  change in pre-ejection period (PEP) during traumatic scripts with VNS compared to sham. PEP is the time from ventricular contraction to aortic valve opening and is a measure of cardiac sympathetic tone
interleukin-6 | baseline
  change in interleukin 6 concentration in blood in response to traumatic scripts with stimulation with VNS versus stimulation with sham

CONTACTS AND LOCATIONS:
Overall Officials: Doug J Bremner, MD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
de identified data will be made available three months after study completion
Supporting Information: Study Protocol, SAP, ICF
Time Frame: three months after study completion
Access Criteria: three months after study completion for twelve months